CLINICAL TRIAL: NCT05627232
Title: A Two-Part Phase 1b Study Evaluating the Combination of Tazemetostat and CPX-351 (Part 1) and Tazemetostat and CPX-351 Following Pre-Treatment With Palbociclib (Part 2) for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Tazemetostat and Palbociclib With CPX-351for R/R AML
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Cohort Closed
Sponsor: Thomas Jefferson University (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22G.769; JT 24252 (Other: JeffTrial Number); 4100095617 (Other Grant/Funding Number: Pennsylvania Department of Health Research Formula CURE)
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tazemetostat; CPX-351; Injections; Daunorubicin; Cytarabine; Liposomes; Biopsy; Specimen Handling; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part I (tazemetostat, CPX-351) (Experimental): Patients receive tazemetostat PO BID on days -1 to 6, and CPX-351 IV over 90 minutes on days 1, 3, and 5. Patients also undergo bone marrow aspiration and biopsy and blood sample collection during screening and on study.
  Interventions: Drug: Tazemetostat; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Biospecimen Collection
- Part II: palbociclib Pre-Treatment Followed by Tazemetostat + CPX-351 (Experimental): Patients receive palbociclib PO QD on days -3 to -1, then tazemetostat PO twice daily (Days -1 to 6), and CPX-351 IV over 90 minutes on days 1, 3, and 5. Patients also undergo bone marrow aspiration and biopsy and blood sample collection during screening and on study.
  Interventions: Drug: Tazemetostat; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Biospecimen Collection; Drug: Palbociclib

INTERVENTIONS:
Drug: Tazemetostat — Given PO
  Other Names: 1403254-99-8; E7438; EPZ-6438; EPZ6438; N-((4,6-Dimethyl-2-oxo-1,2-dihydropyridin-3-yl)methyl)-5-(ethyl(oxan-4-yl)amino)-4-methyl-4'-((morpholin-4-yl)methyl)(1,1'-biphenyl)-3-carboxamide; N-((4,6-dimethyl-2-oxo-1,2-dihydropyridin-3-yl)methyl)-5-(ethyl(tetrahydro-2H-pyran-4-yl)amino)-4-methyl-4'-(morpholinomethyl)-[1,1'-biphenyl]-3-carboxamide
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Palbociclib — Given PO
  Other Names: 571190-30-2; 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991; Pyrido(2,3-d)pyrimidin-7(8H)-one; 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(1-piperazinyl)-2-pyridinyl)amino)-
  Arms: Part II: palbociclib Pre-Treatment Followed by Tazemetostat + CPX-351

SUMMARY:
This is a two-part phase Ib dose escalation study to evaluate the safety and preliminary efficacy of the combination of tazemetostat and CPX-351 following pre-treatment with palbociclib for patients with relapsed or refractory (R/R) acute myeloid leukemia (AML). Part 1 of the study will seek to establish the safety, tolerability, biological activity and recommended Part 2 dose of tazemetostat in combination with standard-dose CPX-351. Once the recommended Part 2 dose is established, the study will proceed to Part 2 where pre-treatment with palbociclib will be administered prior to the tazemetostat/CPX-351 dose combination. The objective of Part 2 is to establish the optimal dose of palbociclib.).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Part 1: To determine the optimal dose of tazemetostat in combination with CPX-351 in patients with R/R-AML.

Part 2: To determine the optimal dose of palbociclib pre-treatment prior to combination of tazemetostat/CPX-351 in patients with R/R-AML.

SECONDARY OBJECTIVE:

I. To evaluate the preliminary efficacy of tazemetostat in combination with CPX-351 (Part 1) and of palbociclib Tazemetostat and Palbociclib with CPX-351for R/R AML pre-treatment prior to tazemetostat/CPX-351 combination (Part 2).

EXPLORATORY OBJECTIVES:

1. To determine whether treatment with the EZH2 inhibitor tazemetostat de-condenses the H3K27me3-marked chromatin of AML blasts.
2. To determine whether cell cycle re-entry of AML cells after palbociclib treatment influences DNA damage and apoptosis induced by combining EZH2 inhibition with anthracycline-based therapy

This is a phase 1, single-institution, two-part, dose-escalation study utilizing tazemetostat in combination with CPX-351 (Part 1) and palbociclib pre-treatment followed by tazemetostat/CPX-351 combination (Part 2) for patients with relapsed or refractory AML who are fit to receive intensive chemotherapy. The study will take place in two parts:

Part 1: Dose escalation via traditional 3+3 design of tazemetostat in combination with CPX-351 .

Part 2: Dose escalation via traditional 3+3 design of palbociclib pre-treatment followed by tazemetostat/CPX-351combination.

After completion of study treatment, patients are followed up at 3 months, 6 months, and 1 year for clinical outcomes including survival.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female >= 18 years of age
* Histologically confirmed acute myeloid leukemia (non-M3) relapsed from or refractory to at least 1 prior line of therapy. Bone marrow aspirate and biopsy within 28 days of screening is acceptable. If no prior bone marrow biopsy is available, bone marrow biopsy must be performed during screening unless:

  * If the subject has >= 20% myeloblasts present in the peripheral blood, a bone marrow biopsy is not necessary to meet this criterion
* Treatment with a prior investigational agent is acceptable so long as it has not been administered within 2 weeks of enrollment and any prior adverse effects have resolved to grade 1 or less with the exception of alopecia
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Life expectancy of at least 4 weeks
* Must be able to consume oral medication
* Subjects must have recovered from the toxic effect of any prior therapy to =< grade 1 (except alopecia)
* Creatine clearance (CrCL) >= 45
* Total bilirubin < 2 x upper limit of normal (ULN)
* Female subjects of childbearing age must have a negative pregnancy test

Exclusion Criteria:

* Subjects with acute promyelocytic leukemia
* Subjects receiving any active chemotherapy agents (except hydroxyurea). Intrathecal methotrexate and cytarabine are permissible
* Subjects whose participation would result in a total cumulative dose of daunorubicin greater than 550 mg/m^2 or greater than 450 mg/m^2 if they previously received mediastinal radiation
* Subjects with evidence of active central nervous system (CNS) leukemia involvement. Lumbar puncture is not required for enrollment in the absence of neurologic symptoms
* Subjects must not be receiving growth factors (except erythropoietin)
* Subjects with currently active second malignancy with the exception of nonmelanoma skin cancer, carcinoma in situ of the cervix, resected prostate cancer with Gleason score =< 6
* Subjects with unstable cardiac disease or uncontrolled arrhythmia
* Subjects with other severe concurrent disease which, in the judgement of the investigator, would make the patient inappropriate to receive high-intensity therapy
* Subjects who are pregnant or breastfeeding
* Subjects with known allergic reactions to components of the study product(s)
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade >= 3 non-hematologic dose limiting toxicities | Up to 1 year
  The primary outcome measure will be grade >= 3 non-hematologic dose limiting toxicities. Adverse events will be coded by organ system and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 5.0. the calculation of adverse events incidences will be passed on number of patients per adverse event category. Standard proportions will be used to report rates of safety endpoints. Summary tables will be presented by dose level, seriousness, severity and relatedness.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 1 year
  Assessment of safety and tolerability: Incidence, nature, and severity of adverse events and incidence, nature and severity of treatment-emergent adverse events. The primary outcome measure will be grade >= 3 non-hematologic dose limiting toxicities. Adverse events will be coded by organ system and graded according to the CTCAE v. 5.0. the calculation of adverse events incidences will be passed on number of patients per adverse event category. Standard proportions will be used to report rates of safety endpoints. Summary tables will be presented by dose level, seriousness, severity and relatedness.
Complete response | Up to 1 year
  Morphologic leukemia-free state: < 5% blasts in bone marrow, no blasts with Auer rods or persistence of extramedullary disease. Morphologic complete response (CR): < 5% blasts in bone marrow with transfusion independence, absolute neutrophil count (ANC) > 1.0 x 10^9/L, platelets >= 100 x10^9/L. CR without minimal residual disease: morphologic CR with negative molecular markers by real-time quantitative polymerase chain reaction or negative multi-parameter flow cytometry. CR with partial hematologic recovery (CRh): as < 5% blasts in bone marrow with no evidence of disease and partial recovery of peripheral blood counts (ANC > 0.5 x 10^9/L and platelets > 50 x 10^9/L). CR with incomplete hematologic recovery (CRi): all CR criteria and transfusion independence but with persistence of neutropenia (ANC < 1.0 x 10^9/L) or thrombocytopenia (platelets < 100 x 10^9/L). Composite complete response: CR + CRh + CRi.
Partial remission (PR) | Up to 1 year
  PR is defined as decrease of at least 50% in the percentage of bone marrow blasts to 5% - 25% and normalization of blood counts.
Relapse | Up to 1 year
  Relapse is defined as reappearance of leukemic blasts in the peripheral blood or > 5% blasts in the bone marrow not attributable to other cause (e.g., bone marrow regeneration after chemotherapy) or extramedullary relapse.
Induction failure/refractory acute myeloid leukemia (AML) | Up to 1 year
  Induction failure/refractory AML defined as failure to attain CR or CRi.
Time to blood count recovery | The number of days until ANC > 1.0 x 10^9/L and platelets >= 100 x 10^9/L from day 1 of treatment, assessed up to 1 year
  95% confidence intervals will be calculated using Kaplan-Meier method.
Relapse free survival | The time measured in months to relapse from day 1 of treatment, assessed up to 1 year
  95% confidence intervals will be calculated using Kaplan-Meier method.
Overall survival | The time measured in months from day 1 of treatment, assessed up to 1 year
  95% confidence intervals will be calculated using Kaplan-Meier method.
Rate of allogeneic stem cell transplantation | Up to 1 year
  Defined as the proportion of patients who undergo allogeneic stem cell transplantation during the study period.
Time to transplant | The time measured in months to allogeneic stem cell transplantation from day 1 of treatment, assessed up to 1 year
  95% confidence intervals will be calculated using Kaplan-Meier method.

OTHER OUTCOMES:
Deoxyribonucleic acid (DNA) damage and apoptosis | Up to day 5
  DNA damage (analysis of gammaH2AX-positive AML cells by confocal microscopy) and apoptosis (Annexin V and caspase 3 activation) will be assessed in S phase-enriched AML cells (16-24 hours post palbociclib treatment) following treatment with the EZH2 inhibitor tazemetostat to de-condense the H3K27me3-marked chromatin and chemotherapy (CPX-351) to induce DNA damage (double strand breaks).

CONTACTS AND LOCATIONS:
Overall Officials: Gina Keiffer, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States